CLINICAL TRIAL: NCT02416713
Title: Way to Safety: Cellphone Blocking Technology to Reduce Cellphone Use While Driving Among Teens
Brief Title: Way to Safety Cellphone Blocking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-11234
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-07

CONDITIONS: Teen Drivers; Motor Vehicle Accident
Keywords: Driving; Teens; Texting; Cellphone; DriveID; Motor vehicle accident

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Education Only (Control) (Placebo Comparator): The Cellcontrol DriveID device will run completely in the background with no observable changes to cellphone functions while driving. During Week Four, participants will be presented educational materials on the dangers of distracted driving.
  Interventions: Other: Education Only
- Opt-in Blocking (Experimental): Participants will have to initiate Cellcontrol DriveID device when entering the vehicle; the blocking settings will be pre-set to block all calls and text messages when the car is in motion.
  Interventions: Device: Cellcontrol DriveID
- Opt-out Blocking (Experimental): Cellcontrol DriveID device will automatically turn on when the teen begins driving and will be pre-set to block all calls and text messages when the car is in motion.
  Interventions: Device: Cellcontrol DriveID
- Opt-out Blocking with Notification (Experimental): Cellcontrol DriveID device will automatically turn on when the teen begins driving and will be pre-set to block all calls and text messages when the car is in motion. If a participant overrides the blocking function, an email will be sent to a parent/guardian.
  Interventions: Device: Cellcontrol DriveID

INTERVENTIONS:
Device: Cellcontrol DriveID — Technology that blocks incoming and outgoing calls and texts.
  Other Names: DriveID
  Arms: Opt-in Blocking; Opt-out Blocking; Opt-out Blocking with Notification
Other: Education Only — No active intervention, educational materials will be provided
  Other Names: Control
  Arms: Education Only (Control)

SUMMARY:
Research participants will be recruited to take part in a randomized control trial. Participants' cellphone use will be observed during an initial baseline period. Participants will then be randomly assigned to one of four conditions: education only (control), opt-in blocking, opt-out blocking, and opt-out blocking with parental notification.

DETAILED DESCRIPTION:
Motor vehicle crashes are the leading cause of death in teens in the United State and for drivers aged 15-19 involved in fatal crashes, 21% of distracted drivers were distracted by the use of cellphones. Nearly 90% of teens expect a response to a text message within 5 minutes, and the compulsion to respond is stronger for messages from close social contacts. This suggests that behavioral-economic interventions such as immediate and frequent incentives are needed to offset the disutility caused by not being able to communicate by cellphone while driving. If proven to be effective, incentives could be scaled up via auto insurance discount contributions, school programs, and parental contributions.

ELIGIBILITY:
Inclusion Criteria:

1. High school student
2. 16 or 17 at start of the study
3. Have a valid driver's license
4. Lives in parent's/guardian's home
5. Drives to school
6. Primarily drive one car
7. Has their own iPhone 4S or newer or Android 4.3 or newer smartphone with data plan
8. Parent/guardian is willing to assist with installation
9. Admit to texting while driving >1 time in the last 30 days

Exclusion Criteria:

1. Already uses a smartphone app or hardware device to limit cellphone use while driving

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine McDonald, PhD, RN, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education Only (Control) | Opt-in Blocking | Opt-out Blocking | Opt-out Blocking With Notification
Started | 8 | 9 | 8 | 10
Completed | 8 | 9 | 8 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education Only (Control) | Opt-in Blocking | Opt-out Blocking | Opt-out Blocking With Notification | Total
Number analyzed (Participants) | 8 | 9 | 8 | 10 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 9 | 8 | 10 | 35
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 6 | 25
  Male | 2 | 2 | 2 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 9 | 8 | 9 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 6 | 7 | 8 | 9 | 30
  More than one race | 1 | 1 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 9 | 8 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Cellphone Unlocks
Description: Change in number of phone unlocks per hour of drive time between intervention period (last 3 weeks) vs. baseline period (last 3 weeks)
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: Phone unlocks per hour
Arm/Group | Education Only (Control) | Opt-in Blocking | Opt-out Blocking | Opt-out Blocking With Notification
Number analyzed (Participants) | 8 | 9 | 8 | 10
Phone unlocks per hour | 0.26 [-0.52 to 1.04] | 0.52 [-0.28 to 1.33] | -0.95 [-3.68 to 1.79] | 1.08 [-1.62 to 3.78]
Statistical Analysis 1: Comparison: Education Only (Control) vs Opt-in Blocking; Test type: Superiority; p = 0.12, Mixed Models Analysis; relative change from baseline = 0.66, 95% CI 2-sided [-0.18 to 1.51]
Statistical Analysis 2: Comparison: Education Only (Control) vs Opt-out Blocking; Test type: Superiority; p = 0.49, Mixed Models Analysis; relative change from baseline = -0.30, 95% CI 2-sided [-1.17 to 0.57]
Statistical Analysis 3: Comparison: Education Only (Control) vs Opt-out Blocking With Notification; Test type: Superiority; p = 0.70, Mixed Models Analysis; Slope = -0.16, 95% CI 2-sided [-1.00 to 0.69]

ADVERSE EVENTS:
Time Frame: 8 weeks (results analysis only uses data from last 3 weeks from baseline and last three weeks from the intervention period)
Arm/Group | Education Only (Control) | Opt-in Blocking | Opt-out Blocking | Opt-out Blocking With Notification
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT02416713/Prot_SAP_000.pdf